CLINICAL TRIAL: NCT04577235
Title: Evaluation of the Correlation Between Thoracic Ultrasound and Thorax Computed Tomography Scores of Patients With Severe COVID 19 Pneumonia in Intensive Care.
Brief Title: Correlation Between Thoracic Ultrasound and Thorax Computed Tomography Scores.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Ayşe Vahapoglu, M.D. Anaesthesiology and Reanimation, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AyşeV
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: COVID-19 Pneumonia; Critical Care; Lung ultrasound; Computed tomography
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Survivors group (Experimental): Lung ultrasound score and computed tomography score were evaluated in the surviving group
  Interventions: Other: severity of lung involvement with COVID-19.
- Non survivors group (Experimental): Lung ultrasound score and computed tomography score were evaluated in the non surviving group
  Interventions: Other: severity of lung involvement with COVID-19.

INTERVENTIONS:
Other: severity of lung involvement with COVID-19. — transthoracic lung ultrasound and throcic CT

SUMMARY:
Coronavirus Disease 19 (COVID-19) pandemic has become a global health problem in a short time due to high infection rate and increasing mortality. Since it is not possible to perform thorax computed tomography (CT) and transfer of patients with COVID-19 pneumonia who are followed up in intensive care, diagnosis and follow-up by lung ultrasound (LUS) is a great advantage nowadays.The investigators aimed to evaluate the correlation between thoracic CT score and LUS score and to determine its relationship with mortality.

Patients who were admitted to intensive care with the diagnosis of COVID-19 pneumonia, who had an initial thorax CT examination and who underwent LUS during admission to the intensive care unit were included in the study. The demographic characteristics, clinical parameters, prognosis, thorax CT and LUS scores of the patients were recorded prospectively. The characteristics of the survived patients and the patients who died were compared.

DETAILED DESCRIPTION:
Thorax CT scoring was performed by an experienced radiologist, while LUS scoring was performed an experienced anaesthesia and reanimation specialist. The demographic characteristics, clinical parameters, prognosis, thorax CT and LUS scores of the patients were recorded prospectively. The correlation between thorax CT score and LUS score was evaluated.Lung ultrasound score (LUSS):

LUS was performed by an intensive care specialist with experience in this field using a 2- to 5-MHz transducer (Esaote MyLabSeven, Getz Healthcare Malaysia). The transducer was covered with a probe cover, and the transducer and ultrasound device were cleaned with disinfectant wipes after each use. LUS examinations were performed at the bedside, in the supine position, and twelve-zone examinations were performed. Each hemithorax is separated into 6 quadrants: anterior, lateral, and posterior zones (separated by the anterior and posterior axillary lines) each divided in upper and lower portion (Figure 1). Each zone was scored according to the LUS pattern as follows: the presence of lung sliding with A-lines or fewer than two isolated B-lines, scored 0; when multiple well-defined B-lines presented, scored 1; the presence of multiple coalescent B-lines, scored 2; and when presented with a tissue pattern characterized by dynamic air bronchograms (lung consolidation), scored 3. The worst ultrasound pattern observed in each zone was recorded and used to calculate the sum of the scores (total score = 36).

CT Technique and Image Interpretation The thorax CT scans in the study were obtained using the low dose protocol of our hospital with a 128-slice multi-detector CT scanner (Optima; General Electric Healthcare, Wisconsin, USA). All CT scans were performed during a single breath-hold without contrast administration.

As in the ultrasound evaluation, each lung was divided into anterior, lateral and posterior quadrants based on the anterior and posterior axillary lines, and then each quadrant was divided into upper and lower sections. Each quadrant was scored between 0-3. It was scored 0 when there was no parenchymal involvement, 1score when the parenchymal involvement rate was between 0 and 33%, 2 score when it was between 33% and 66%, and 3score when it was above 66%.

ELIGIBILITY:
Inclusion criteria:

* Over 18 years of age

Exclusion criteria:

* Under 18 years of age
* Previous lung resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
The evaluation of the correlation between the baseline LUS score and mortality rate of patients with severe COVID-19 pneumonia who were followed up in the intensive care unit | 2 month
  LUS score

SECONDARY OUTCOMES:
The evaluation of the correlation between the baseline CT score and mortality rate of patients with severe COVID-19 pneumonia who were followed up in the intensive care unit | 2 month
  CT skore

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Taksim Research and Education Hospital, Istanbul, Gazi̇osmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No